CLINICAL TRIAL: NCT03803072
Title: A Novel Diet Approach to Combat Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/2271
Record Dates: First submitted 2018-12-18; First posted 2019-01-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Diabetes, Gestational
Keywords: Exercise therapy; Diet; Prevention and control
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (TRE) (Experimental): prolonging the duration of fasting between the last evening meal and the first meal of the next day
  Interventions: Behavioral: time restricted eating (TRE)
- control (No Intervention): Standard care. Will receive a booklet about physical activity recommendations and healthy eating in pregnancy

INTERVENTIONS:
Behavioral: time restricted eating (TRE) — Participants will attend a face-to-face meeting with the researchers at the last day of the first week of data collection (habitual diet and physical activity period) where they will be counselled to consume all food and fluid within a 8-10 h time window of their choice starting no later than 09.00 h for five weeks. During the intervention period, they will be counselled by weekly phone calls to provide encouragement, support and monitoring to improve adherence to the TRE window.
  Arms: Time restricted eating (TRE)

SUMMARY:
There is an urgent need to implement novel diet approaches to combat the increasing rates of gestational diabetes mellitus (GDM). The primary aim of this study is to establish the feasibility of time-restricted eating in pregnancy, to prepare for future larger controlled trials in this research project to determine the efficacy of time-restricted eating in women at risk of GDM. Expectations:

1. Women who have an increased risk of GDM will be able to adhere to time reduced eating during pregnancy.
2. Time reduced eating will improve short-term glycemic control in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* carrying one singleton live foetus
* in pregnancy week 12-30
* having at least one risk factor for gestational diabetes mellitus (GDM) according to Norwegian guidelines for GDM screening: pre-pregnancy BMI > 25 kg/m2, GDM in previous pregnancy, primiparae aged > 25 years, first degree relative with diabetes mellitus, Asian or African ethnicity, previous delivery of new-born > 4.5 kg
* understand written and spoken Norwegian language

Exclusion Criteria:

* habitual eating window < 12 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in average time-window for energy intake | Change between baseline (pre-intervention) time-window for energy intake to average time-window for energy intake during the 5-week intervention period
  Average daily time-window for energy intake will be registered through log books.
Weekly adherence rates for time restricted eating (TRE) | Weekly measures throughout the 5 week period of TRE intervention
  The number of days per week that the participants are able to adhere to TRE, as calculated as weekly average of days with a time-window ≤ 10 hours

SECONDARY OUTCOMES:
Perceived barriers to the protocol assessed with an unstructured interview | Weekly phone calls to participants in TRE group during the 5-week intervention period and after 6 weeks
  Participants will be asked about which barriers they perceived as challenging regarding keeping to a TRE schedule and if they have strategies to overcome these barriers.
Subjective appetite sensations assessed by Visual Analogue Scales | Once weekly throughout 6 weeks, on a weekday.
  Paper line scales 100 mm on scales for Hunger ("How hungry are you": From "Not at all" = 0 on the scale to "Extremely. As hungry as I have ever felt" =100 on the scale, Fullness (From "Not at all" = 0 on the scale to "Extremely. As full as I have ever felt" = 100 on the scale, Satiety ("How satiated are you" From "Not at all" =0 on the scale to "Extremely" =100 on the scale, Desire to eat ("How strong is your desire to eat" From "Very weak. Extremely low" = 0 on the scale to "Very strong. Extremely high" = 100 on the scale and Prospective consumption (quantity) ("How much do you think you could (or would want to) eat right now?" From "Nothing at all" = 0 on the scale to "A very large amount" = 100 on the scale. Scales will be filled in in the morning, before dinner and at bedtime.
Change between baseline and post-intervention in fasting glucose | 6 weeks
  Post-intervention fasting glucose minus pre-intervention fasting glucose
Change between baseline and post-intervention in postprandial glucose | 6 weeks
  Blood glucose levels 120 minutes after ingestion of 75 g glucose (oral glucose tolerance test)
Change between baseline and post-intervention in fasting insulin | 6 weeks
  Circulating insulin levels
Change between baseline and post-intervention in postprandial insulin | 6 weeks
  Circulating insulin levels 120 minutes after ingestion of 75 g glucose.
Change between baseline and post-intervention blood pressure | 6 weeks
  Diastolic and systolic blood pressure
Change between baseline and post-intervention body mass | 6 weeks
  Body mass in kg.
Change in total cholesterol | 6 weeks
  Total cholesterol measured in blood
Change in triglycerides | 6 weeks
  Triglycerides measured in blood
Change in HDL cholesterol | 6 weeks
  HDL cholesterol measured in blood
Change in LDL cholesterol | 6 weeks
  LDL cholesterol measured in blood
Change in HbA1c | 6 weeks
  HbA1c measured in blood
Continuous glucose monitoring | 6 weeks
  Interstitial glucose measurements
Change between baseline and post-intervention fat mass | 6 weeks
  Fat mass in kg and percent of body mass
Change between baseline and post-intervention muscle mass | 6 weeks
  Muscle mass in kg
Change between baseline and post-intervention visceral fat area | 6 weeks
  Visceral fat area in squared cm.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — Department of circulation and medical imaging, NTNU
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No